CLINICAL TRIAL: NCT06881745
Title: NUTRI_ACTIVE Study: Lifestyle and Nutrition Evaluation in Physically Active People and Athletes
Brief Title: Lifestyle and Nutrition Evaluation in Physically Active People and Athletes
Acronym: NUTRI_ACTIVE
Status: Recruiting | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: 65268/2023
Record Dates: First submitted 2024-08-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Dietary Habits; Nutritional Status; Body Composition; Athlete
Keywords: Mediterranean Diet; Physical Activity; Athletes; Nutritional status; Nutrition knowledge
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the dietary intake, nutrition knowledge and body composition in Italian athletes and physically active adults. This is a nonprofit study aimed at improving clinical practice. The main questions it aims to answer are:

* Assessment of level of adherence to Mediterranean Diet using MEDI-LITE questionnaire
* Assessment of nutrition knowledge
* Current dietary intake and eating habits evaluation and comparison to the recommendations, according to sport practised
* Eating behaviour assessment

Participants will undergo the following assessments: anthropometric and body composition assessments, Resting Metabolic Rate measurement, Dietary intake assessment, Nutrition knowledge, Lifestyle and behaviour, Physical activity assessment.

DETAILED DESCRIPTION:
Participants will undergo the following assessments:

1) Baseline assessment Nutrition assessment will be performed at the Laboratory of Nutrition Education and Sports Nutrition of the Department of Public Health, Experimental and Forensic Medicine at the University of Pavia.

The preliminary classification of the participants includes an evaluation of the inclusion and exclusion criteria of the study. The participants will be classified according to the type of sport practised (team sports, endurance/long distance, middle distance/power, speed/strength, precision, racquet sports, combat/weight-making). Professionals from the research team involved in the research project will carry out this selection and classification.

All variables will be reported at study baseline. Preliminar general information will be collected (age, gender, educational level, occupation, lifestyle, weight history, nutrition intervention in the past…).

All participants will be fully evaluated by a trained team using the standardised procedure:

* weight, height measurement
* waist, hip, arm circumference
* skinfold thickness at the biceps, triceps, subscapular, suprailiac, abdominal, pectoral, mid-axillary, thigh sites

Body composition evaluation using the Bioelectrical Impedance Analysis, which is a non-invasive and commonly used method for assessing body composition (BIA 101 BIVA PROTM- AKERN). It works by passing a low-level electrical current through the body and measuring the resistance encountered by the current. Body tissues with different compositions (such as muscle, fat, and bone) conduct electricity differently, allowing BIA to estimate the proportion of lean body mass and body fat.

Resting Metabolic Rate measurement will be done with Indirect calorimetry that is the gold standard method to assess the Resting Metabolic Rate (RMR). This instrument will be used to measure RMR in the morning, in a fasted, rested state. The indirect calorimetry method requires the subject to wear a mask connected with a respiratory gas analyser. The duration of the test is about 30 minutes. There are no risks for the patient carrying out this test.

Dietary intake of this sample will be evaluated with a food frequency questionnaire (FFQ) composed of 110 items elaborated by Marventano and colleagues in 2016. The food items on the FFQ are grouped according to their nutrient contents in eight food groups, as follows: (a) Meat and fish products; (b) Sweets, nuts and snacks; (c) Vegetables; (d) Fruits; (e) Drinks; (f) Cereals and starchy foods; (g) Milk and dairy products; and (h) Oils and seasonings.

Participants will also complete a 7-day food diary. It records the type and quantity of food and beverages, time and place of consumption, psychological states and social events that interfere in the eating process. Supplement use will also be registered.

Data from the FFQ and food diary will be compared with each participant's nutritional requirements based on measurement of basal metabolic rate by indirect calorimetry adjusted for physical activity level.

Nutrition knowledge will be evaluated with the General and Sport Nutrition Knowledge questionnaire (GeSNK) that is composed by 62 items divided into two main areas which are respectively related to:

* Nutrition Knowledge in general (29 items)
* Sports Nutrition Knowledge (33 items)

Adherence to Mediterranean Diet will be evaluated with a specific tool: Mediterranean Diet Score (MEDI-LITE). The Medi-Lite adherence score consists of 9 items that assess the daily consumption of fruit, vegetables, cereals, meat and meat products, dairy products, alcohol, and olive oil, and the weekly consumption of legumes and fish. For each food group, there are three categories of consumption, based on data available in the literature in relation to adherence to the Mediterranean diet and health status. The final score is obtained from the sum of all these scores, and it ranges from 0 (low adherence) to 18 (high adherence).

Teruel Orthorexia Scale (TOS) will be also administered to participants. It is validated in Italy. It is a 17-item self-report measure articulated in 2 subscales: healthy orthorexia (9 items), which indicates a healthy, nonpathological interest in proper nutrition, and orthorexia nervosa (8 items), which represents an extreme preoccupation with healthy diet that may lead to relevant emotional, social, and cognitive impairments. All items are rated on a 4-point Likert scale, ranging from 0 (completely disagree) to 3 (completely agree).

Eating Attitude Test (EAT-26): it is the most widely used test to measure the symptoms and concerns characteristic of eating disorders. Scores greater than 20 indicate a need for further investigation by a qualified professional. Low scores (below 20) can still be consistent with serious eating problems, as denial of symptoms can be a problem with eating disorders. Results should be interpreted along with weight history, current BMI (body mass index), and percentage of Ideal Body Weight.

Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.

International Physical Activity Questionnaires (IPAQ) - long form will also be administered to the participants. IPAQ was developed in the late 1990s as an instrument for cross-national assessment of duration and frequency of physical activity in the last seven days. This questionnaire analyses five domains: a) job-related activity; b) transportation; c) housework, house maintenance, caring for family d) recreation, sport and leisure time e) time spent sitting. This tool can be useful for the general lifestyle assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old and ≤ 65 years old
* Regular physical activity (at least 150 minutes of moderate-intensity aerobic physical activity; or at least 75 of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week)
* All genders

Exclusion Criteria:

* Sedentary population: < 150 minutes of moderate-intensity aerobic physical activity or < 75 minutes of vigorous-intensity aerobic physical activity throughout the week
* Age: < 18 years old and > 65 years old
* Presence of diseases (i.e. diabetes, hypertension, dyslipidemia, metabolic syndrome, neurological diseases,…) and/or injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be composed of volunteers from Pavia city, territorial sport centres, amateur sport clubs and National Sport Federations. The participants will be recruited at the Laboratory of Nutrition Education and Sport Nutrition at University of Pavia who agree to participate in the study and have signed the relevant informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of level of adherence to Mediterranean Diet | Baseline
  Adherence to Mediterranean Diet will be evaluated with Mediterranean Diet Score (MEDI-LITE). that consists of 9 items that assess the daily consumption of fruit, vegetables, cereals, meat and meat products, dairy products, alcohol, and olive oil, and the weekly consumption of legumes and fish. For each food group, there are three categories of consumption, based on data available in the literature in relation to adherence to the Mediterranean diet and health status. The final score is obtained from the sum of all these scores, and it ranges from 0 (low adherence) to 18 (high adherence).

SECONDARY OUTCOMES:
Assessment of nutrition knowledge | Baseline
  Nutrition knowledge will be evaluated with the General and Sport Nutrition Knowledge questionnaire (GeSNK) that is composed by 62 items divided into two main areas which are respectively related to:
  Nutrition Knowledge in general (29 items) Sports Nutrition Knowledge (33 items)
Current dietary intake and eating habits evaluation and comparison to the recommendations, according to sport practised | Baseline
  Dietary intake will be evaluated with a food frequency questionnaire (FFQ) composed of 110 items. The food items on the FFQ are grouped according to their nutrient contents in eight food groups, as follows: (a) Meat and fish products; (b) Sweets, nuts and snacks; (c) Vegetables; (d) Fruits; (e) Drinks; (f) Cereals and starchy foods; (g) Milk and dairy products; and (h) Oils and seasonings.
  Participants will also complete a 7-day food diary. It records the type and quantity of food and beverages, time and place of consumption, psychological states and social events that interfere in the eating process. Supplement use will also be registered.
  Data from the FFQ and food diary will be compared with each participant's nutritional requirements based on measurement of basal metabolic rate by indirect calorimetry adjusted for physical activity level.
Eating behaviour assessment | Baseline
  Eating behavior will be assessed with two principle questionnaires:
  Teruel Orthorexia Scale (TOS), a 17-item self-report measure articulated in 2 subscales: healthy orthorexia (9 items), which indicates a healthy, nonpathological interest in proper nutrition, and orthorexia nervosa (8 items), which represents an extreme preoccupation with healthy diet that may lead to relevant emotional, social, and cognitive impairments. All items are rated on a 4-point Likert scale, ranging from 0 (completely disagree) to 3 (completely agree).
Eating behavior assessment | Baseline
  Eating Attitude Test (EAT-26) will be used to measure the symptoms and concerns characteristic of eating disorders. Scores greater than 20 indicate a need for further investigation by a qualified professional. Scores below 20 can still be consistent with serious eating problems, as denial of symptoms can be a problem with eating disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Ferraris, PhD, Principal Investigator — University of Pavia
Locations (1):
- Laboratory of Food Education and Sport Nutrition, Department of Public Health, Experimental and Forensic Medicine, University of Pavia, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: web site of Laboratory of Food Education and Sport Nutrition — https://spmsf.dip.unipv.it/it/ricerca/laboratori-e-strumentazione/laboratorio-di-educazione-alimentare-e-nutrizione-sportiva